CLINICAL TRIAL: NCT02511496
Title: Status of Chronic Liver Disease in Hepatitis C Virus (HCV) Patients Coinfected With Human Immunodeficiency Virus (HIV) in Andalusia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: HEP-COI-1-2014
Record Dates: First submitted 2015-03-11; First posted 2015-07-30 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Hepatitis C; Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Hepatitis C, Chronic; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the current situation and follow-up of chronic hepatitis C virus (HCV) infection in patients co-infected with human immunodeficiency virus (HIV) in Andalusia.

DETAILED DESCRIPTION:
In subjects co-infected with HIV, treatment of chronic HCV infection is particularly complex and requires considerable resources, including a very high cost is likely to increase with new antivirals.

A precise knowledge of the situation in each hospital would facilitate adequate provision of personal and material resources needed to adequately address this disease in each center and in the Community as a whole. Because all or the vast majority of patients coinfected HIV / HCV are staffed by specialists who are part of Hepavir group and / or Sociedad Andaluza de Enfermedades Infecciosas (SAEI), they are ideal for carrying out this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 with HIV infection and active chronic hepatitis or SVR after treatment.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample consists of all HIV-infected patients co-infected with an active chronic HCV.
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sustained virological response | Up to twelve months
  This variable will be collected as follow at each clinical visit: i) yes; ii) not valuable (patients still on treatment); or, iii) no (patients who has not initiated treatment in the corresponding visit).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Rivero Juárez, Principal Investigator — Instituto Maimónides de Investigación Biomédica de Córdoba (IMIBIC)

REFERENCES:
- [Derived] Rivero-Juarez A, Guijo-Rubio D, Tellez F, Palacios R, Merino D, Macias J, Fernandez JC, Gutierrez PA, Rivero A, Hervas-Martinez C. Using machine learning methods to determine a typology of patients with HIV-HCV infection to be treated with antivirals. PLoS One. 2020 Jan 10;15(1):e0227188. doi: 10.1371/journal.pone.0227188. eCollection 2020. PMID 31923277